CLINICAL TRIAL: NCT01215968
Title: A Study to Evaluate the Effect of LY2189265 on Gastric Emptying Using Scintigraphy in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of LY2189265 on the Speed at Which Food and Drink Leaves the Stomach in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13598; 2009-017305-11 (EudraCT Number); H9X-EW-GBDM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Each participant will receive placebo on Week 1. Participants randomized to placebo will receive once-weekly doses of placebo on Weeks 2 to 5.
  Placebo will be administered by single subcutaneous injection into the skin of the abdominal wall.
  Participants regularly taking metformin will continue their normal dosing regimen throughout the study.
  Interventions: Drug: Placebo
- LY2189265 (Experimental): Participants randomized to LY2189265 will receive once-weekly doses of LY2189265 on Weeks 2 to 5.
  1.5 milligram (mg) LY2189265 will be administered by single subcutaneous injection into the skin of the abdominal wall.
  Participants regularly taking metformin will continue their normal dosing regimen throughout the study.
  Interventions: Biological: LY2189265; Drug: Placebo

INTERVENTIONS:
Biological: LY2189265 — 1.5 mg administered subcutaneously
  Arms: LY2189265
Drug: Placebo — Administered subcutaneously

SUMMARY:
The primary purpose of this Study is to help answer the following research question(s).

* How does LY2189265 affect gastric emptying (the speed at which food and drink leaves the stomach) in patients with Type 2 diabetes?
* How does LY2189265 affect how the body handles metformin (a drug used to treat Type 2 diabetes)?
* Is LY2189265 safe and are any side effects associated with it?

The study will be participant-blind in Week 1, and participant- and investigator-blind from Week 2 through Week 5.

Each participant will receive placebo on Week 1 and once-weekly doses of LY2189265 or Placebo on Weeks 2 to 5. Participants taking metformin for the treatment of Type 2 Diabetes Mellitus (T2DM) will continue taking metformin as part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are males or females, diagnosed with Type 2 Diabetes Mellitus for greater than or equal to 3 months prior to screening.
2. Male patients agree to use a reliable method of birth control during the study and for 3 months following the last dose of study drug. Female patients must be of non-child-bearing potential due to surgical sterilization or menopause.
3. Have a body mass index (BMI) between 18.5 and 40.0 kilogram/square meter (kg/m²), inclusive.
4. Have Type 2 Diabetes Mellitus controlled with diet and exercise alone or are stable on a single oral antidiabetic medication (e.g. metformin) prior to screening, and have been taking a stable dose for >7 days prior to the first dosing occasion.
5. Have a fasting blood glucose value at screening >126 milligram/deciliter (mg/dL) (7.0 [millimoles/liter] mmol/L) for patients on a controlled diet, and >108 mg/dL (6.0 mmol/L) for patients on oral antidiabetic medication, with an upper limit of 180 mg/dL (approximately 9.9 mmol/L) in each case.
6. Have a hemoglobin A1c (HbA1c) (indicates what your average blood glucose level has been in the past 3 months) value at screening (or within 4 weeks prior to screening) of 6.5% to 9.5%. If HbA1c is between 6.1% and 6.5%, patients may participate in the study providing they are receiving permissible oral antidiabetic medication.
7. Have clinical laboratory test results within normal ranges as determined by the study doctor.
8. Can provide enough blood in order to undergo the blood sampling required for the study.
9. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
10. Have signed the consent form approved by Lilly and the Ethical Review Board (ERB) governing the site.

    Exclusion Criteria:
11. Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
12. Have previously been exposed to, or have known allergies to glucagon-like-peptide-1 (GLP-1)-related compounds including LY2189265.
13. Are persons who have previously completed or withdrawn from this study or any other study investigating LY2189265 or have received glucagon-like peptides or incretin mimetics in the past 3 months.
14. Have taken certain Type 2 Diabetes medications within 30 days prior to screening.
15. Have an abnormality in the electrocardiogram (ECG) performed at screening.
16. Have poorly controlled high blood pressure (systolic blood pressure >160 millimeters of mercury [mmHg] and/or diastolic blood pressure >100 mmHg).
17. Have a history or presence of respiratory, liver, kidney, hormonal, blood, or neurological disorders which may put the patient at risk when taking the study medication; or may interfere with the interpretation of data.
18. Have a history or presence of cardiovascular disorder within the last year, or signs of congestive heart failure, or are expected to require coronary artery bypass surgery or angioplasty.
19. Have a history or presence of pancreatitis or certain gastrointestinal disorders.
20. Have been exposed to radiation from clinical trials and from diagnostic X-ray or are exposed routinely via your job worker.
21. Have any non-removable metal objects such as metal plates, screws etc. in their chest or abdominal area.
22. Have had acute diarrhea or constipation within 14 days of study screening.
23. Show evidence of significant active neuropsychiatric disease.
24. Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
25. Intend to start new medication during the study, including over-the-counter and herbal medication.
26. Have donated blood of more than 500 milliliter (mL) within the last month prior to screening.
27. Have an average weekly alcohol intake that exceeds the study centre's guidelines and are unwilling to adhere to the alcohol restrictions in place throughout the study.
28. Smoke more than 10 cigarettes (or equivalent in nicotine) per day, and are unwilling to stop smoking on the day of medication administration or are unable to abide by clinical research unit (CRU) restrictions on other inpatient days.
29. Are allergic to eggs or other components of the meals to be served.
30. Are patients who, in the opinion of the investigator, are in any way unsuitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo on Week 1 and once-weekly doses of placebo on Weeks 2 to 5.
- LY2189265: Participants received placebo on Week 1 and once-weekly doses of 1.5 milligram (mg) LY2189265 on Weeks 2 to 5.
Period: Overall Study
Arm/Group | Placebo | LY2189265
Started | 13 | 25
Received at Least 1 Dose of Study Drug | 13 | 24 (25 participants received placebo during Week 1.)
Completed | 11 | 18
Not Completed | 2 | 7
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 2 | 4
Not completed — Not received study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY2189265 | Total
Number analyzed (Participants) | 13 | 25 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (14.0) | 58.9 (9.8) | 56.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 11 | 20 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 25 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 24 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 25 | 38

OUTCOME MEASURES:

1. Primary Outcome: Time Required for 50% of Radioactivity To Be Emptied From the Stomach by Scintigraphy
Description: After at least 8 hours fasting, participants received a radiolabeled breakfast containing technetium-99m-tin colloid (99mTc-tin colloid). After which serial anterior and posterior scintigraphy images were taken. Data presented are the time required for 50% of radioactivity to be emptied from stomach. The results presented are Geometric Least Squares (LS) Mean. LS Mean values were controlled for weeks.
Time Frame: Days 3, 10,17, 24 and 31
Population: All randomized participants who received study drug, a radiolabeled breakfast, and had scintigraphy images taken. Those who violated protocol were excluded.
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Placebo | LY2189265
Number analyzed (Participants) | 10 | 15
hours
  Day 3 | 1.44 [1.22 to 1.69] | 1.72 [1.43 to 2.06]
  Day 10 | 1.41 [1.20 to 1.66] | 3.77 [3.15 to 4.51]
  Day 17 (n=9, 14) | 1.60 [1.36 to 1.89] | 3.32 [2.76 to 4.00]
  Day 24 (n=9, 14) | 1.47 [1.25 to 1.73] | 3.28 [2.72 to 3.94]
  Day 31 (n=10, 13) | 1.46 [1.24 to 1.71] | 3.15 [2.61 to 3.81]
Statistical Analysis 1: Comparison: LY2189265; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio is the Geometric LS Means of Day 10 over Day 3; Ratio of Geometric LS Mean = 2.19, 90% CI 2-sided [1.83 to 2.62]
Statistical Analysis 2: Comparison: LY2189265; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio is the Geometric LS Means of Day 17 over Day 3; Ratio of Geometric LS Mean = 1.94, 90% CI 2-sided [1.61 to 2.33]
Statistical Analysis 3: Comparison: LY2189265; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio is the Geometric LS Means of Day 24 over Day 3; Ratio of Geometric LS Mean = 1.91, 90% CI 2-sided [1.59 to 2.29]
Statistical Analysis 4: Comparison: LY2189265; Test type: Superiority or Other; Mixed Linear effects model analyses; Ratio is the Geometric LS Means of Day 31 over Day 3; Ratio of Geometric LS Mean = 1.84, 90% CI 2-sided [1.52 to 2.22]

2. Secondary Outcome: Area Under the Curve (AUC) of Metformin
Description: Metformin was used as a secondary marker in the study to correlate the effect of LY2189265 on gastric emptying to the pharmacokinetics (PK) (measured as AUC) of concomitant medications. Participants taking metformin for treatment of Type 2 Diabetes Mellitus (T2DM) underwent PK assessments for metformin in parallel to their scintigraphy assessments for gastric emptying. AUC of metformin was calculated during one dosing interval.
Time Frame: Days 3, 17 and 31
Population: All randomized participants who received both study drug and immediate release metformin, and had PK data. Those who violated protocol were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Placebo | LY2189265
Number analyzed (Participants) | 6 | 12
nanograms*hour/milliliter (ng*h/mL)
  Day 3 | 13600 (49) [11228 to 16824] | 13700 (40)
  Day 17 | 14600 (47) [12523 to 18766] | 15300 (43)
  Day 31 (n=6, 11) | 14600 (47) [12941 to 19429] | 15800 (43)

3. Secondary Outcome: Maximum Concentration (Cmax) of Metformin
Description: Metformin was used as a secondary marker in the study to correlate the effect of LY2189265 on gastric emptying to the pharmacokinetics (PK) (measured as Cmax) of concomitant medications. Participants taking metformin for treatment of Type 2 Diabetes Mellitus (T2DM) underwent PK assessments for metformin in parallel to their scintigraphy assessments for gastric emptying.
Time Frame: Days 3, 17 and 31
Population: All randomized participants who received both study drug and immediate release metformin, and had pharmacokinetic (PK) data. Those who violated protocol were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Placebo | LY2189265
Number analyzed (Participants) | 6 | 12
nanograms/milliliter (ng/mL)
  Day 3 | 1610 (48) | 1690 (47)
  Day 17 | 1690 (48) | 1500 (53)
  Day 31 (n=6, 11) | 1770 (46) | 1680 (44)

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of Metformin
Description: Metformin was used as a secondary marker in the study to correlate the effect of LY2189265 on gastric emptying to the pharmacokinetics (PK) (measured as Tmax) of concomitant medications. Participants taking metformin for treatment of Type 2 Diabetes Mellitus (T2DM) underwent PK assessments for metformin in parallel to their scintigraphy assessments for gastric emptying.
Time Frame: Days 3, 17 and 31
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Placebo | LY2189265
Number analyzed (Participants) | 6 | 12
hour
  Day 3 | 1.00 [1.00 to 2.03] | 2.02 [1.00 to 4.10]
  Day 17 | 2.02 [1.02 to 8.00] | 2.05 [0.96 to 4.02]
  Day 31 (n=6, 11) | 1.53 [0.98 to 4.00] | 2.02 [1.00 to 4.03]

5. Secondary Outcome: Number of Participants With Clinically Significant Effects
Description: Adverse events (AEs) were considered clinically significant effects. A summary of serious adverse events (SAEs) and other nonserious AEs are located in the Reported Adverse Event section.
Time Frame: Baseline through 5 weeks
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo (Week 1): Participants received placebo on Week 1 and went on to receive once-weekly doses of 1.5 milligram (mg) LY2189265 on Weeks 2 to 5.
- LY2189265: Participants received placebo on Week 1 and once-weekly doses of 1.5 mg LY2189265 on Weeks 2 to 5.
Arm/Group | Placebo | Placebo (Week 1) | LY2189265
Number analyzed (Participants) | 13 | 25 | 24
participants
  SAEs | 0 | 0 | 0
  Other nonserious AEs | 7 | 11 | 20

ADVERSE EVENTS:
Arm/Group | Placebo | Placebo (Week 1) | LY2189265
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 7/13 | 11/25 | 20/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Placebo (Week 1) (N=25) | LY2189265 (N=24)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (8)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (19)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 7 (18)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (6)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 12 (25)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (11)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 2 (2) | 2 (4)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (5) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 8 (12)
Increased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (5)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (3) | 4 (4) | 5 (7)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days